CLINICAL TRIAL: NCT02839928
Title: Nasal Ketamine: Mild Sedation and Analgesia for Minor Procedures in the Pediatric Emergency Department (ED)
Brief Title: Nasal Ketamine for Minor Procedures in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0034-16-KMC
Record Dates: First submitted 2016-07-13; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ketamine; Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): The experimental arm consists of children given intranasal Ketamine 1 mg/kg, once
  Interventions: Drug: Intranasal ketamine; Device: Intranasal atomizer; Drug: EMLA

INTERVENTIONS:
Drug: Intranasal ketamine — The experimental arm consists of an single intranasal administration of Ketamine (Ketalar).
  Other Names: Ketalar
Device: Intranasal atomizer — Ketamine will be applied to each nare via intranasal atomizer
  Other Names: LMA MAD intranasal atomizer
Drug: EMLA
  Other Names: EMLA cream, a topical analgesic, will be applied prior to the procedure

SUMMARY:
Nasal Ketamine has previously been tested in children for deep sedation or preoperative anxiolysis. The investigators intend to test the efficacy of low dose nasal Ketamine in children undergoing minor procedures in the emergency department.

DETAILED DESCRIPTION:
The investigators propose a feasibility study of intranasal ketamine to provide analgesia and anxiolysis before minor procedures. This will be a single-blinded randomized study of inhaled ketamine in a convenience sample of children ages 4-12 years of age undergoing minor procedures. For the purpose of this study, the investigators will limit minor procedures to venipuncture and IV placement, and will further limit the patient population to children who are deemed by the investigators to show resistance to IV placement or venipuncture without premedication. The investigators have chosen the ages 4-12 years because these children are verbal and able to rate their pain on the VAS scales, because they are likely to require restraint and to require a staff member to assist parents with restraint, and because the Green study found this age range to have the fewest adverse events with ketamine.

The investigators propose a uniform dosing of 50 mg/ml intranasal ketamine at 1 mg/kg. Ketamine will be diluted to achieve volumes between 0.5-1 ml distributed between nares. The plasma concentration of intranasal ketamine is just over a fifth of IV ketamine, and the peak serum concentration is reached an average of fifteen minutes later than IV ketamine. Thus, intranasal administration found to have achieved mild sedation at 1 mg/kg would be expected to achieve a lower level of sedation than a 0.2 mg/kg slow IV administration, which is compatible with subdissociative dosing used for analgesia. A 1 mg/kg intranasal dose is also consistent with the lower end of the dosing spectrum used in the anesthesia literature for preoperative sedation.

The investigators propose a pilot study of 20 children ages 4-12 years undergoing venipuncture or IV insertion. After obtaining informed consent from a single parent (the investigators request exclusion from requiring consent from both parents), the children will be assigned to receive 1 mg/kg intranasal ketamine via atomizer. Consent will occur after the treating physician has decided that the child requires bloodwork or IV placement, and will not impact this decision.

All children will receive EMLA. EMLA cream is the standard of care in our area and we feel that it would not be ethical to withhold EMLA for the purpose of the study. Ketamine will add to the incomplete analgesia of EMLA, and may be a better option than EMLA in children who are known to have difficult venous access. EMLA is not universally effective -- having been found to decrease VAS pain scores by only 61%-- and causes vasoconstriction, which can increase the procedural fail rate.

Ketamine will be administered 30 minutes after EMLA is applied. At or about the 45 minute mark, the procedure will be attempted.

All children will receive continuous monitoring of pulse oximetry, blood pressure and pulse rate from the time medication is administered until the child is discharged from the emergency department. All children will be under the direct and continuous observation of ED staff. The procedure will be completed within twenty minutes of the completion of the nasal administration.

After the procedure is completed, children will be asked to rate the level of procedural pain on the Faces scale. A parent and the nurse at the procedure will rate the estimated procedural pain on the VAS scale. Child, parent as nurse will be blinded to each other's score.

The investigators intend to show that nasal ketamine requires a minimal disruption in ED resources and treatment time, effectively treats pain and increases the child's compliance with venipuncture and IV placement, increases parent satisfaction, and is without serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Children age 4-12 years old presenting to the pediatric ED
* Children determined by the treating physician to require either venipuncture or IV placement
* Children determined by the treating physician to show resistance to the procedure without pre-medication

Exclusion Criteria

* ASA 3 or higher
* Weight below 15 kg or above 50 kg
* Hypoxia below 95% on presentation or noted to be tachypneic for age or dyspneic.
* Judged by staff to need an urgent procedure that cannot be delayed (i.e. Nursing triage levels 1-2)
* An existing source of pain that results in a VAS greater than 3 at triage (i.e. Headache, fracture)
* More than four prior ED visits in the last four months
* Developmentally delayed and unable to reliably rate pain

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pain score (VAS) | Up to 24 weeks
  The investigators will record the visual analog scale pain score as reported by patients and caregivers both before and after the administration of intranasal ketamine

CONTACTS AND LOCATIONS:
Overall Officials: Eric Scheier, MD, Principal Investigator — Physician, pediatric emergency department

IPD SHARING:
Plan to Share IPD: No